CLINICAL TRIAL: NCT00523250
Title: A Phase II, First-in-human Dose-escalation, Double-masked, Randomized, Vehicle-controlled, Dose-response Study Assessing the Safety and Ocular Hypotensive Efficacy of AR-102 in Subjects With Elevated Intraocular Pressure
Brief Title: Ocular Hypotensive Efficacy of AR-102
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR102-CS201
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- AR-102 0.003% Ophthalmic Solution (Experimental): q.d. ocular
  Interventions: Drug: AR-102 0.003% Ophthalmic Solution
- AR-102 0.005% Ophthalmic Solution (Experimental): q.d. ocular
  Interventions: Drug: AR-102 0.005% Ophthalmic Solution
- AR-102 0.01% Ophthalmic Solution (Experimental): q.d. ocular
  Interventions: Drug: AR-102 0.01% Ophthalmic Solution
- AR-102 0.03% Ophthalmic Solution (Experimental): q.d. ocular
  Interventions: Drug: AR-102 0.03% Ophthalmic Solution
- AR-102 Vehicle Ophthalmic Solution (Experimental): q.d. ocular
  Interventions: Drug: AR-102 Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: AR-102 0.003% Ophthalmic Solution
  Arms: AR-102 0.003% Ophthalmic Solution
Drug: AR-102 0.005% Ophthalmic Solution
  Arms: AR-102 0.005% Ophthalmic Solution
Drug: AR-102 0.01% Ophthalmic Solution
  Arms: AR-102 0.01% Ophthalmic Solution
Drug: AR-102 0.03% Ophthalmic Solution
  Arms: AR-102 0.03% Ophthalmic Solution
Drug: AR-102 Vehicle Ophthalmic Solution
  Arms: AR-102 Vehicle Ophthalmic Solution

SUMMARY:
A double-masked, randomized, vehicle-controlled, dose-response study assessing the safety and ocular hypotensive efficacy of AR-102 in subjects with elevated intraocular pressure. The Null hypothesis is that the ocular hypotensive efficacy of each dose of AR-102 Ophthalmic Solution will not be different from that of its vehicle.

DETAILED DESCRIPTION:
A double-masked, randomized, vehicle-controlled, dose-response study assessing the safety and ocular hypotensive efficacy of AR-102 in subjects with elevated intraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater (male, or female not of childbearing potential).
* Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT) in the study eye(s).
* Corrected visual acuity by ETDRS in each eye of +1.0 logMAR units or better

Exclusion Criteria:

* Known hypersensitivity to any component of the formulation or to topical anesthetics
* Previous glaucoma intraocular surgery or laser procedures in study eye(s)
* Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, cardiovascular or endocrine disorders) which might interfere with the study.
* Participation in any study involving an investigational drug within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be mean change from baseline in intraocular pressure at each time point. | One week

SECONDARY OUTCOMES:
The primary safety endpoints will be visual acuity, objective biomicroscopic and ophthalmoscopic examination, and subjective comfort as measured by adverse events in response to subject questionnaires | One week

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Van Haarlem, MD, Study Director — Aerie Pharmaceuticals, Inc.
Locations (8):
- United States (8):
  - Soilsh Practice, Pasadena, California
  - Bacharach practice, Petaluma, California
  - Hernando Eye Institute, Brooksville, Florida
  - Taustine Eye Center, Louisville, Kentucky
  - Mundorf Practice, Charlotte, North Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Texan Eye, Austin, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas